CLINICAL TRIAL: NCT04503330
Title: Using Buccal Mucosal Graft as an Augmention Graft for Complex Cases of Iatrogenic Pelviureteric Junction Obstruction and Long Segment Ureteric Stricture Disease.
Brief Title: Buccal Mucosal Graft for the Repair of Iatrogenic Pelviureteric Junction Obstruction or Ureteric Stricture.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abozamel, principal investigator urologist, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cairo univeristy
Record Dates: First submitted 2020-08-03; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Pelvi Ureteric Junction Obstruction or Ureteral Stricture
MeSH Terms: conditions — Multicystic renal dysplasia, bilateral

STUDY DESIGN:
Intervention Model Description: 20 patients with iatrogenic pelviureteric junction obstruction or ureteric stricture disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with iatrogenic PUJO (Experimental): patients with iatrogenic PUJO or long segment ureteric stricture disease for safety and efficacy of using buccal graft for repair
  Interventions: Procedure: buccal mucosal graft to repair iatrogenic PUJO

INTERVENTIONS:
Procedure: buccal mucosal graft to repair iatrogenic PUJO — Augmented buccal mucosal graft anastomosis to repair iatrogenic PUJO or long segment ureteric stricture disease

SUMMARY:
Prospective study to evaluate the safety and efficacy of using buccal mucosal graft for repairing complex cases of iatrogenic pelvi ureteric junction obstruction and long segment ureteric stricture disease.

DETAILED DESCRIPTION:
A graft of buccal mucosa will be used to augment either the narrow unhealthy pelviureteric junction or a narrow long segment of the ureter.

after freeing the narrowed part, a posterior incision will be made in the ureter or renal pelvis then the graft will be implanted on the psoas muscle using interrupted sutures in a position the allows easy anastomosis to the ureter or renal pelvis.

Alternatively a lateral incision in the renal pelvis or the ureter may be done for the graft anastomosis and then surrounded with omenal flap to ensure a good blood supply for the graft.

ELIGIBILITY:
Inclusion Criteria:

- any patient with iatrogenic pelviureteric junction obstruction or long segment ureteric stricture

Exclusion Criteria:

* elderly patients unfit for general anaesthesia.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with patent renal pelvis and ureter after surgery. | 3 months
  3 months after surgery Diuretic renography will be done to judge patency of the pelvis and ureter and resolution of hydronephrosis

IPD SHARING:
Plan to Share IPD: Yes
study protocol statistical analysis results
Supporting Information: Study Protocol, SAP
Time Frame: June 2021
Access Criteria: through clinical trials webpage